CLINICAL TRIAL: NCT05077111
Title: A Comparative Study Between Thoracic Epidural Anesthesia in Non-Intubated Video-Assisted Thoracoscopes and the Conventional General Anesthesia With One Lung Ventilation
Brief Title: A Comparative Study Between Regional Anesthesia in Thoracoscopes and the Conventional General Anesthesia
Acronym: VATS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mohamed Reda Ashour (Other)
Responsible Party: Sponsor-Investigator, Mohamed Reda Ashour, Assistant lecturer, Dept of Anesthesia, Intensive Care and Pain Management, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FMASU M D 389/2019
Record Dates: First submitted 2021-09-19; First posted 2021-10-14 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-09

CONDITIONS: Pleural Effusion, Malignant; Pleural Mesothelioma; Pleural Empyema; Pulmonary Diseases or Conditions; Pleural Neoplasms; Pulmonary Atelectasis; Pleural Diseases; Pericardial Effusion; Mediastinal Lymphadenopathy; Pneumothorax and Air Leak; Hemothorax; Pyopneumothorax
Keywords: thoracocentesis,; pleural, biopsy, wash, effusion,; ventilation; thoracic epidural; non intubated VATS,; pericardiocenthesis
MeSH Terms: conditions — Pleural Effusion, Malignant; Mesothelioma, Malignant; Empyema, Pleural; Lung Diseases; Pleural Neoplasms; Pulmonary Atelectasis; Pleural Diseases; Pericardial Effusion; Pneumothorax; Hemothorax; Respiratory Aspiration | interventions — Anesthesia, General; One-Lung Ventilation

STUDY DESIGN:
Intervention Model Description: the study will include 40 participants, randomized into 2 equal groups, Group A: Awake participants will receive sole Thoracic Epidural Anesthesia. Group B: Participants receiving General Anesthesia with One Lung Ventilation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): sole Thoracic Epidural Anesthesia
  Interventions: Procedure: Thoracic Epidural Anesthesia
- Group B (Active Comparator): General Anesthesia with One Lung Ventilation
  Interventions: Procedure: General Anesthesia with One Lung Ventilation

INTERVENTIONS:
Procedure: Thoracic Epidural Anesthesia — Group A pre-medicated once using Midazolam 3-4mg intravenous (IV) and Fentanyl 50mcg, placed in the setting position. Using a winged 18G (Gadge), 9cm length Tuohy Epidural needle, a 20G springwound closed tip epidural catheter be inserted between T3-T4. A test dose (5ml) 2% Lidocaine given, followed by 5-8 ml Bupivacaine 0.5% and 50mcg Fentanyl as a loading dose. Further top-up dose of 5 ml Bupivicaine 0.5% after 45 minutes.
  Arms: Group A
Procedure: General Anesthesia with One Lung Ventilation — Group B premedicated once by 3-4mg Midazolam IV, Ranitidine 50mg, Metoclopramide 10mg and Dexamethasone 4mg. Preoxygenation with 100% O2. Induction of anesthesia with Propofol (2mg/kg) and Fentanyl (1mcg/kg). Tracheal intubation by 37-39 Fr Double Lumen Endotracheal Tube insertion facilitated with Cisatracurium 0.1mg/kg. and confirmation of its position by Fiberoptic Bronchoscopy. Selective Lung Ventilation strategy can be performed through the endobroncheal tube of the non operated lung once needed. Anesthesia maintained with Isoflurane (1-2%) and Cisatracurium (0.05mg/kg per dose). Later, anesthesia discontinued and extubation after full neuromuscular recovery after reversal of muscle relaxant by Neostigmine (0.05mg/kg) and Atropine (0.02mg/kg).
  Arms: Group B

SUMMARY:
Video-assisted thoracic surgery (VATS) is usually performed with general anesthesia and single lung ventilation. However, performing thoracic surgery under awake regional anesthesia has several potential advantages including avoidance of airway trauma and ventilator dependence associated with endotracheal intubation, besides promoting enhanced recovery after surgery and shorter mean hospital stay.

DETAILED DESCRIPTION:
The aim of this study is to investigate the feasibility and the effect of Thoracic Epidural Anaesthesia for awake thoracic surgery to speed up recovery in patients as well as avoiding the complications accompanying General Anesthesia with one lung ventilation.

Type of Study: Prospective randomized clinical study. Study Setting: This study will be conducted in Ain Shams University Hospitals..

Study Period: Expected for two years starting from 2019.

Sampling Method: Randomized sampling by a computer generated random numbers table.

Sample Size: 40 patients. Sample size was calculated using PASS 11 program for sample size calculation and according to the (Pompeo et al., 2004) study, the mean PaO2 perioperatively in the awake group = -3±1.5 mmHg and in the second group = -6.5±1.83 mmHg. Sample size of 40 cases per group (total 40) can detect this difference with power 100% and α-error 0.05.

ELIGIBILITY:
Inclusion Criteria:

* ASA less than or equal II.
* The procedure expected to be completed within 2 hours.

Exclusion Criteria:

* Patients with expected difficult airway management.

  * Hemodynamically unstable patients.
  * Persistent cough or high airway secretions.
  * Severe Emphysema or clinical signs of active infectious disease.
  * Hypoxemia (PaO2 <60 mmHg) or hypercarbia (PCO2 >50 mmHg)
  * Coagulopathy (INR >1.5).
  * Obesity (BMI >30 Kg/m 2 ).
  * Infection at the injection site, allergy to local anesthetics.
  * Neurological disorders: seizures, intracranial mass or brain edema.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-01-15 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-10-15 (Estimated)

PRIMARY OUTCOMES:
Perioperative changes in blood gases | Imediately before operation, intraoperatively per hour, and postoperatively till 24 hours
  Ratio of arterial oxygen tension to fraction of inspired oxygen (PaO2/FiO2), arterial carbon dioxide tension (PaCO2). Hypoxemia is defined as peripheral oxygen saturation (SpO2) < 92% on room air with a need for oxygen supplementation.

SECONDARY OUTCOMES:
Postoperative pain | Postoperatively at 3,12 and 24 hours
  The Visual Analogue Scale (VAS) consists of a 10 cm straight line with the endpoints defining extreme limits of "no pain at all" (0 cm) and "pain as bad as it could be" (10 cm). The patient is asked to mark his pain level on the line between the two endpoints. The distance between 0 and the mark then defines the subject pain score.
Postoperative opioid needs | Postoperatively during the 24 hours after regaining sensation
  Pethidine consumption
Hospital stay | from day of operation to discharge; average, 5 days
Perioperative changes in heart rate | Immediately before the operation, intraoperatively per hour, and postoperatively till 24 hours
  heart rate (HR) in beats per minute (bpm)
The onset of ambulance. | During the 24 hours after regaining of full motor power
  Rate of occurence of falling after ambulance will be recorded in each group.
Number of episodes of Post Operative Nausea and Vomiting (PONV) | During the 24 hours postoperatively
Perioperative changes in mean arterial pressure | Immediately before the operation, intraoperatively per hour, and postoperatively till 24 hours
  mean arterial pressure (MAP) in mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Samia A M Abdel Latif, Professor, Study Chair — Department of Anesthesia, Intensive care and pain management, Ain Shams University.; Waleed El Taher, Professor, Study Director — Department of Anesthesia, Intensive care and pain management, Ain Shams University.; Hany H El Sayed, Professor, Study Director — Department of Thoracic Surgery, Ain Shams University.; Ahmed F Koraitim, MD, Study Director — Department of Anesthesia, Intensive care and pain management, Ain Shams University.; Mohamed A A alhadidy, MD, Study Director — Department of Anesthesia, Intensive care and pain management, Ain Shams University.
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: starting 6 months after publication

REFERENCES:
- [Background] Chen KC, Cheng YJ, Hung MH, Tseng YD, Chen JS. Nonintubated thoracoscopic lung resection: a 3-year experience with 285 cases in a single institution. J Thorac Dis. 2012 Aug;4(4):347-51. doi: 10.3978/j.issn.2072-1439.2012.08.07. PMID 22934136
- [Background] Deng HY, Zhu ZJ, Wang YC, Wang WP, Ni PZ, Chen LQ. Non-intubated video-assisted thoracoscopic surgery under loco-regional anaesthesia for thoracic surgery: a meta-analysis. Interact Cardiovasc Thorac Surg. 2016 Jul;23(1):31-40. doi: 10.1093/icvts/ivw055. Epub 2016 Mar 16. PMID 26984963
- [Background] Pompeo E, Mineo D, Rogliani P, Sabato AF, Mineo TC. Feasibility and results of awake thoracoscopic resection of solitary pulmonary nodules. Ann Thorac Surg. 2004 Nov;78(5):1761-8. doi: 10.1016/j.athoracsur.2004.05.083. PMID 15511470
- [Background] Pompeo E, Sorge R, Akopov A, Congregado M, Grodzki T; ESTS Non-intubated Thoracic Surgery Working Group. Non-intubated thoracic surgery-A survey from the European Society of Thoracic Surgeons. Ann Transl Med. 2015 Mar;3(3):37. doi: 10.3978/j.issn.2305-5839.2015.01.34. PMID 25815298
- See also: May awake video-assisted thoracoscopic surgery with thoracic epidural anesthesia use routinely for minimaly invasive thoracic surgery procedures in the future? — https://www.ijsurgery.com/index.php/isj/article/view/2746

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-12-17): https://cdn.clinicaltrials.gov/large-docs/11/NCT05077111/Prot_SAP_000.pdf
  • Informed Consent Form (2019-12-17): https://cdn.clinicaltrials.gov/large-docs/11/NCT05077111/ICF_001.pdf